CLINICAL TRIAL: NCT02295358
Title: The Effect of Omega-3 Fatty Acid Supplementation on Intraocular Pressure & Ocular Surface
Status: Withdrawn | Type: Observational
Why Stopped: Project never got initiated
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0235
Record Dates: First submitted 2014-11-13; First posted 2014-11-20 (Estimated); Last update posted 2015-07-09 (Estimated); Status verified 2015-07

CONDITIONS: Open Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed with the intention to further elucidate the effects of omega-3 fatty acids on intraocular pressure (IOP) and signs/symptoms of dry eye. Prior studies have shown statistically significant lowering of IOP with use of omega-3 fatty acids but have only been performed in animal models. This study will be the first to attempt replication in human models. A limited number of studies have shown an increase in tear production/volume as well as a decrease in the subjective symptoms of dry eye, but more studies are needed to better define these effects. Better understanding of the effects of this supplement on intraocular pressure and dry eye will contribute to the expanding knowledge about the pathophysiology of glaucoma/ocular hypertension and dry eye syndrome and potentially lead to further studies about new potential treatment options for these conditions.

DETAILED DESCRIPTION:
The purpose of this research project is to determine the effects of omega-3 fatty acid supplementation on intraocular pressure (IOP) as well as the signs and symptoms of dry eye. We hypothesize that dietary omega-3 fatty acid supplementation will be associated with a significant change in intraocular pressure compared to baseline measurements prior to beginning supplementation. We further hypothesize that omega-3 fatty acid supplementation will be associated with a significant increase in tear production and volume as well as a significant change in patients' subjective complaints of dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Ocular Hypertension or Open Angle Glaucoma of mild to moderate severity, with or without previously diagnosed dry eye syndrome, who are currently on monotherapy with a prostaglandin analog.
* Age 40-89 of either gender, of any race/ethnicity

Exclusion Criteria:

* Females who are currently pregnant or planning to become pregnant during the study period
* Age <40 years old
* Diagnosis of any other form of glaucoma other than open-angle
* Patients with known hypersensitivity (i.e., anaphylactic reaction) to omega-3 fatty acids or any of its components
* Patients with cirrhosis or with known liver disease
* Patients with diagnosed celiac disease
* Patients with a hypersensitivity to fish or shellfish
* Patients with paroxysmal or persistent atrial fibrillation
* Patients who are currently using medical or recreational marijuana
* Patients currently on any anticoagulation therapy including warfarin, dabigatran, apixaban, rivaroxaban, clopidogrel, cilostazol, dipyridamole, prasugrel, ticlopidine, ticagrelor
* Patients currently on Lovaza, an omega- 3 fatty acid supplement requiring a prescription
* Patients with any recent ocular surgery or laser treatment within 3 months

Ages: 40 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosis of Ocular Hypertension or Open Angle Glaucoma of mild to moderate severity, with or without previously diagnosed dry eye syndrome, who are currently on monotherapy with a prostaglandin analog. Age 40-89 of either gender, of any race/ethnicity
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
The Effect of Omega-3 Fatty Acid Supplementation on Intraocular Pressure | Change in intraocular pressure from baseline over 3 month
  Intraocular pressure is measured at the study start, and after three month on supplementation.

SECONDARY OUTCOMES:
The Effect of Omega-3 Fatty Acid Supplementation on Ocular Surface | Change in Ocular Surface from baseline over 3 month
  Tear breakup time, corneal fluorescein staining, and tear osmolarity of Ocular Surface is measured at the study start, and after three month on supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Leonard K Seibold, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Eye Center, Aurora, Colorado, United States